CLINICAL TRIAL: NCT01074177
Title: Understanding Mechanisms of Acquired Resistance to BIBW2992
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Texas (Other); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Lecia V. Sequist, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-092
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer; EGFR Mutations
Keywords: BIBW 2992; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIBW 2992 (Experimental): BIBW 2992 Taken orally once a day
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — Taken orally once a day
  Other Names: Afatinib

SUMMARY:
In this research study we are looking to see how effective BIBW 2992 is at suppressing the development of the T790M mutation in non-small cell lung cancer (NSCLC) patients. Epidermal growth factor receptors (EGFR) are proteins found on the surface of some cancer cells that promote a growth signal. Some cancer drugs for NSCLC work to block this signal from reaching its target on the cancer cells which in turn may slow or stop the cancer from growing. However, many times patients with EGFR mutations will stop responding to these cancer drugs and develop drug-resistance because they have developed a specific EGFR mutation called T790M. BIBW 2992 may prevent the T790M mutation from becoming active and therefore slow disease progression.

DETAILED DESCRIPTION:
* Participants will take tablets of BIBW 2992 once a day during each cycle. Each cycle is 28 days (4 weeks).
* Participants will come to the clinic on Day 1, 8 and 15 of Cycle 1. For Cycle 2 through 8, they will need to come to the clinic on Day 1. After Cycle 8, they will have study visits every 2 months.
* The following tests and procedures will be performed at these clinic visits: physical examination, routine blood tests, research blood samples, EKG (every fourth cycle starting cycle 5), ECHO or MUGA (every fourth cycle starting cycle 5), an assessment of the tumor by CT or MRI scan (every 8 weeks).
* Participants may continue to participate in this research study as long as their tumor does not grow and their disease does not worsen and they do not have any severe side effects.
* Participants will have a tumor biopsy performed at the end of their participation in this study if their tumor is growing or if they have a new tumor. The purpose of this biopsy is to assess for the presence or the absence of the mutation T790M.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed stage IIIB, IV or recurrent non-small cell lung cancer
* A somatic mutation in epidermal growth factor receptor (EGFR) must be present as documented by a CLIA-certified laboratory
* There must be radiographic measurable or evaluable disease
* Participants must be willing, at the time of signing consent, to agree to a future biopsy of their tumor tissue at the time of disease progression, provided such a biopsy is safe and feasible at that time.
* Performance status must be 0, 1 or 2 on the Eastern Cooperative Oncology Group scale
* 18 years of age or older
* Normal organ and marrow function as outlined in the protocol
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Prior EGFR tyrosine kinase inhibitor therapy (including gefitinib, erlotinib, or any experimental EGFR TKI agents)
* Known brain metastases, unless they have undergone definitive therapy and are neurologically stable at the time of study entry
* Standard chemotherapy or radiation less than 2 weeks of starting BIBW 2992, or experimental systemic cancer therapy less then 4 weeks of starting BIBW 2992. Note that prior palliative radiation to bony disease, CNS disease, or a limited thoracic area is allowed if there is measurable or progressive disease outside the field of radiation.
* Another malignancy within the last 3 years (except for non-melanoma skin cancer or a non-invasive/in situ cancer)
* Known pre-existing and clinically active interstitial lung disease
* Significant gastrointestinal disorders with diarrhea as a major symptom
* History of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia, or myocardial infarction within 6 months
* Cardiac left ventricular function with resting ejection fraction <50%
* Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the study drug
* Pregnancy or breast feeding
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of BIBW 2992
* Life expectancy of < 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia V. Sequist, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BIBW 2992
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BIBW 2992
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
Brain Metastasis Present [Count of Participants; unit: Participants]
  Yes | 11
  No | 13
Prior Chemotherapy [Count of Participants; unit: Participants]
  Yes | 6
  No | 18
EGFR Mutation [Count of Participants; unit: Participants] — The specific mutation that occurred in the gene for Epidermal Growth Factor Receptor (EGFR)
  Participants
    Exon 19 deletion | 10
    L858R | 8
    Exon 20 insertion | 3
    G719A | 2
    S768I | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Have a T790M Mutation on Their Progression Biopsy.
Time Frame: At the time of disease progression (median duration of 11.4 months from start of treatment)
Population: The 14 participants that experienced disease progression and were also eligible to be biopsied.
Measure: Count of Participants; unit: Participants
Arm/Group | BIBW 2992
Number analyzed (Participants) | 14
Participants | 4

2. Secondary Outcome: Response Rate
Description: The number of participants with either a complete response (CR) or partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
  * CR: Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm
  * PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline and then after the end of every two 28 day cycles until treatment is discontinued; median duration of followup of 19.3 months
Measure: Number; unit: participants
Arm/Group | BIBW 2992
Number analyzed (Participants) | 24
participants
  Complete Response | 0
  Partial Response | 14

3. Secondary Outcome: Median Progression-free and Overall Survival
Description: The progression-free and overall survival times. Overall survival is measured from the start of treatment until the time of death or until the participant is lost to follow-up. Progression free survival is measured from the start of treatment until the time of progression, death, or until the participant is lost to follow-up (whichever occurs first). Progression is defined as having at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study with at least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions denotes disease progression.
Time Frame: start of treatment, at the time of disease progression, time of death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BIBW 2992
Number analyzed (Participants) | 24
Months
  Progression Free Survival | 11.4 [5.9 to 13.7]
  Overall Survival | 20.8 [15.1 to 40.5]

4. Secondary Outcome: Number of Participants With Biopsy Complications From Repeat Tumor Biopsies
Description: The number of participants with biopsy complications from repeat tumor biopsies taken following disease progression. Biopsy complications are any adverse events considered to be potentially related to the biopsy.
Time Frame: 7 days post biopsy and ≥ 30 days post-biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | BIBW 2992
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after last dose was received. Treatment continued until the participant had disease progression, experienced unacceptable toxicity, died, was lost to follow-up, or until the physician decided it was in their best interest to stop treatment (median duration of approximately 11 months).
Arm/Group | BIBW 2992
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIBW 2992 (N=24)
INR Increased (Investigations) | 1 (1)
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIBW 2992 (N=24)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 4 (13)
Hypertension (Vascular disorders) | 3 (3)
Fatigue (General disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 9 (19)
Weight loss (Investigations) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (13)
Nail changes (Skin and subcutaneous tissue disorders) | 5 (6)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Skin-other (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 20 (45)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 3 (3)
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 8 (8)
Taste disturbance (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 2 (2)
GI-other (Gastrointestinal disorders) | 8 (10)
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 13 (16)
Infection Gr0-2 neut, skin (Infections and infestations) | 2 (2)
Infection Gr0-2 neut, ungual (Infections and infestations) | 3 (3)
Infection Gr0-2 neut, upper airway (Infections and infestations) | 2 (3)
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 2 (2)
Infection Gr0-2 neut, vagina (Infections and infestations) | 6 (8)
Alkaline phosphatase (Investigations) | 7 (7)
ALT, SGPT (Investigations) | 3 (7)
AST, SGOT (Investigations) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Creatinine (Investigations) | 7 (27)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Investigations) | 3 (3)
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 12 (16)
Neurologic-other (Nervous system disorders) | 6 (15)
Dry eye syndrome (Eye disorders) | 4 (4)
Abdomen, pain (Gastrointestinal disorders) | 6 (7)
Back, pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest wall, pain (General disorders) | 11 (19)
Chest/thoracic pain NOS (General disorders) | 3 (3)
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Head/headache (Nervous system disorders) | 21 (40)
Joint, pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Renal/GU-other (Renal and urinary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT01074177/Prot_SAP_000.pdf